CLINICAL TRIAL: NCT06247358
Title: Assessment of Frailty, Physical Capacity and Lung Function in Postoperative Cardiac Surgery Patients: an Observational and Prospective Clinical Study
Brief Title: Frailty, Physical Capacity and Lung Function in Postoperative Cardiac Surgery Patients
Status: Recruiting | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Rafael M. Ianotti, PT, Clinical Research Coordinator - Physiotherapy Division - Heart Institute (InCor), University of Sao Paulo General Hospital
Other Study IDs: CAAEE: 73168923.7.0000.0068
Record Dates: First submitted 2023-12-19; First posted 2024-02-07 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-03

CONDITIONS: Cardiac Infarct; Cardiac Valve Disease; Fragility; Physical Disability
Keywords: Cardiac surgery; Short Physical Performance Battery; 1-minute sit-tostand test; Spirometry; muscular strength
MeSH Terms: conditions — Myocardial Infarction; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational and prospective study is to investigate changes in physical performance, lung function, and respiratory and peripheral muscle strength in patients during the postoperative period following coronary artery bypass grafting (CABG) and valve replacement surgery..

DETAILED DESCRIPTION:
This study aims to investigate the physical changes in patients undergoing myocardial revascularization surgery and valve replacement. It will observe alterations in physical performance, lung function, and muscle strength during the postoperative period. The study, observational and prospective, will include individuals aged ≥18 scheduled for these surgeries, evaluating them preoperatively, post-intensive care unit discharge, and before hospital discharge. Assessments involve tests like the Short Physical Performance Battery, 1-minute sit-to-stand test, Clinical Frailty Scale, manovacuometry, dynamometry, and spirometry to identify frailty and measure muscle and lung function. The study also aims to explore predictive variables for functional loss and mortality during hospitalization.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years
* Both genders
* Elective coronary artery bypass grafting surgery
* Elective Heart valve surgery
* Absence of cognitive or peripheral motor impairment that prevents the performance of functional tests in the preoperative period.

Exclusion Criteria:

* Surgeries performed via lateral thoracotomy or minithoracotomy
* Reoperation for any reason
* Presence of cognitive or peripheral motor impairment that prevents the performance of functional tests in the postoperative period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the preoperative period of elective coronary artery bypass grafting and valve replacement surgery
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
To investigate changes in physical performance measured by Short Physical Performance Battery (SPPB) | Baseline (one day before the surgery), after the surgery (the day immediately after ICU discharge) and through study completion, an average of 15 days.
  Measures: walking speed, standing balance and sit-to-stand performance.
To investigate changes in physical performance measured by Six-Minute Walk Test. | Baseline (one day before the surgery), after the surgery (the day immediately after ICU discharge) and through study completion, an average of 15 days.
  Measures: the assessment will take place in a flat 30-meter corridor, marked every 1 meter with non-slip flooring, and the patient will be instructed to walk for six minutes as fast as possible.
To investigate changes in physical performance by 1-minute sit-to-stand test (1-MSTST) | Baseline (one day before the surgery), after the surgery (the day immediately after ICU discharge) and through study completion, an average of 15 days.
  Measure: number of 1-MSTST repetitions.
To investigate changes in peripheral muscle strength | Baseline (one day before the surgery), after the surgery (the day immediately after ICU discharge) and through study completion, an average of 15 days.
  Measure: hand grip strengh measure (Kgf)
To investigate changes in respiratory muscle strength: | Baseline (one day before the surgery), after the surgery (the day immediately after ICU discharge) and through study completion, an average of 15 days.
  Measures: maximal inspiratory and expiratory pressure (cmH2O)
To investigate changes in lung function test measure by spirometry: | Baseline (one day before the surgery), after the surgery (the day immediately after ICU discharge) and through study completion, an average of 15 days.
  Measures: FVC (L), FEV1 (L), FEF (L/s) and FEF 25-75 (%)
To investigate frailty by Clinical Frailty Scale (CFS) | Baseline (one day before the surgery), after the surgery (the day immediately after ICU discharge) and through study completion, an average of 15 days.
  The minimal value is 1 and the maximal is 9 in which the lowest scores mean worse outcomes.

SECONDARY OUTCOMES:
To explore potential preoperative and immediate postoperative risk factors as predictors of functional loss. | Baseline (one day before the surgery) during the immediate postoperative period.
  Occurrence of comorbidities and clinical variables associated with functional decline
To investigate hemodynamic behavior during the Short Physical Performance Battery (SPPB). | Immediately before and after the SPPB.
  Measures: heart rate, systolic blood pressure, diastolic blood pressure and mean arterial pressure.
To investigate hemodynamic behavior during the 1-minute sit-to-stand test (1-MSTST). | Immediately before and after the 1-MSTST tests.
  Measures: heart rate, systolic blood pressure, diastolic blood pressure and mean arterial pressure.
To investigate respiratory behavior during the Short Physical Performance Battery (SPPB). | Immediately before and after the SPPB.
  Measures: respiratory rate, Borg dyspnea scale and peripheral oxygen saturation.
To investigate respiratory behavior during 1-minute sit-to-stand test (1-1-MSTST). | Immediately before and after the 1-MSTST tests.
  Measures: respiratory rate, Borg dyspnea scale and peripheral oxygen saturation.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael M Ianotti, PT, Principal Investigator — Instituto do Coração - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo
Locations (1):
- Instituto do Coração - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil